CLINICAL TRIAL: NCT06344481
Title: A Prospective, Multicenter, Single-Arm, 2-Phase First-in-Human Feasibility Study of the HYALEX® Cartilage System
Brief Title: The Hyalex First-in-Human Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hyalex Orthopaedics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-00003
Record Dates: First submitted 2024-03-21; First posted 2024-04-03 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Cartilage Injury
Keywords: Knee; Cartilage; Lesion
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Hyalex Cartilage System (Experimental): Implantation of Hyalex Cartilage Knee Implant
  Interventions: Device: Surgical (Hyalex Cartilage Knee Implant)

INTERVENTIONS:
Device: Surgical (Hyalex Cartilage Knee Implant) — Implantation of Hyalex Cartilage Knee Implant.

SUMMARY:
The Hyalex First-in-Human Study is a prospective, multicenter, open-label, single-arm, 2-phase, first-in-human study to evaluate the safety and technical performance of the HYALEX Knee Cartilage System for replacement of loss of articular cartilage and bone of the knee femoral condyles in symptomatic patients who require surgical treatment.

ELIGIBILITY:
Inclusion Criteria - Phase 1

1. 21-65 years.
2. Body Mass Index (BMI) ≤ 35.
3. Singular treatable joint surface lesion, ICRS Grade 3 or 4, located on the medial or lateral femoral condyle.
4. Symptomatic, single treatable area 1 - 3.8cm2.
5. Knee Injury and Osteoarthritis Outcome Score (KOOS) pain subscale score between 20 and 65.
6. Stable knee.
7. Non-responsive to a minimum of 3 weeks of conservative treatment, consisting of non-steroidal anti-inflammatory drugs and/or physical therapy.

Inclusion Criteria - Phase 2

1. 21-65 years.
2. Body Mass Index (BMI) ≤ 35.
3. Up to three treatable joint surface lesion(s), ICRS Grade 3 or 4, located on the medial or lateral femoral condyle(s).
4. Symptomatic total treatable area 1 - 10cm2.
5. Knee Injury and Osteoarthritis Outcome Score (KOOS) pain subscale score between 20 and 65.
6. Stable knee.
7. Non-responsive to a minimum of 3 weeks of conservative treatment, consisting of non-steroidal anti-inflammatory drugs and/or physical therapy.

Exclusion Criteria - Phase 1 & 2

HYALEX Implant, Surgical Technique, and Lesion Site Exclusions:

1. Known allergy to polyurethanes, bone cement, acrylic, or titanium.
2. Lack of 2mm of healthy cartilage (ICRS Grade 0 or 1) and 2mm of vital bone wall on all sides of the implant site.
3. Osteochondral defect affecting subchondral bone more than 11mm in depth from adjacent non-defect articular surface.
4. Bipolar cartilage lesions involving patellar or tibial lesions ICRS Grade 3 - 4 opposite the lesion intended for treatment.
5. Insufficient bone stock or bone density determined intra-operatively preventing implant press fit.

Patient Orthopaedic Health Exclusions:

1. Kellgren and Lawrence (KL) grade 3 or 4 on standing radiographs as defined:
2. Hip-knee-ankle (HKA) angle of greater than +/- 5 degrees (varus or valgus malalignment > 5 degrees) on standing X-ray.
3. Lack of normally functioning contralateral knee that restricts activity.
4. Insufficiency fracture of the femoral condyle or tibial plateau.
5. Recent Osteochondritis Dissecans within 1 year.
6. Diagnosis of a concomitant knee injury which the investigator believes may interfere with study participation or confound effectiveness assessment.
7. Any known systemic cartilage and/or bone disorder, such as but not limited to osteoporosis, chondrodysplasia or osteogenesis imperfecta.
8. A symptomatic musculoskeletal condition in the lower limbs that could impede effectiveness measurements in the target knee.
9. Any known tumor of the treatment knee.
10. Prior radiation therapy to the knee joint.
11. Clinically significant or symptomatic vascular or neurological disorder of the lower extremities affecting gait or function.
12. Untreated ACL and/or PCL deficiency or complex ligamentous instability of the study knee according to IKDC Grade C (abnormal) or D (severely abnormal).

Previous Surgery and Intervention Exclusions:

1. Previous surgery in the past 6 months on the index knee except for:

   1. Diagnostic knee arthroscopy and/or debridement / chondroplasty, and
   2. Meniscectomy
2. Previous intra-articular injections, including HA and steroids, within the last 3 months prior to the date of surgery.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Freedom from implant rejection and infection. | Through 24 months.
  Assess the safety (implant rejection, infection) and tolerability of the Hyalex Cartilage Implant.
Change in the Knee Injury & Osteoarthritis Outcome Score (KOOS) from baseline at 12 months. | Through 12 months.
  The KOOS assesses patient pain, other symptoms, function in daily living, function in sport and recreation, and knee related quality of life. Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Domzalski, MD, Principal Investigator — SPORTO, Łódź, Poland
Locations (2):
- Poland (2):
  - SPORTO, Lodz
  - LIFE Medical Center, Warsaw